CLINICAL TRIAL: NCT03572153
Title: Self-Administered Hypnosis Treatment for the Management of Hot Flashes in Women: A Randomized Clinical Trial
Brief Title: A Mind-Body Intervention for Hot Flash Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Gary R. Elkins, Director of Mind-Body Medicine Research Lab, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1237087; R01AT009384 (NIH); 2018.063 (Other: U-M Rogel Cancer Center Protocol Review Committee); HUM00146427 (Other: U-M Institutional Review Board)
Record Dates: First submitted 2018-06-17; First posted 2018-06-28 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Hot Flashes; Postmenopausal Symptoms; Breast Cancer
Keywords: Hot Flashes; Postmenopausal Symptoms; Hypnotic Relaxation Therapy; Mind Body; Hypnosis
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and either be assigned to the self-hypnosis group or a self-administered white noise hypnosis group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administered Hypnosis (Experimental): Self-administered hypnosis will be practiced daily using different audio recordings using the researcher's voice. Participants will practice hypnosis at home after completing the two study sessions.
  Interventions: Behavioral: Self-Administered Hypnosis
- Self-Administered White Noise Hypnosis (Active Comparator): Self-administered white noise hypnosis will be practiced daily using a white noise recording. Participants will practice hypnosis at home after completing the two consent and education sessions.
  Interventions: Behavioral: Self-Administered White Noise Hypnosis

INTERVENTIONS:
Behavioral: Self-Administered Hypnosis — Participants will be listening to six 20-minute hypnosis audio recordings with hypnotic induction. Participants will be encouraged to practice daily, and each recording will build on the content of the previous recordings. They will also be provided with booklets of information about hot flashes, including treatment options.
  Arms: Self-Administered Hypnosis
Behavioral: Self-Administered White Noise Hypnosis — Participants will be listening to the same 20-minute white noise audio recordings for 6 weeks and will be encouraged to practice daily.They will also be provided with booklets as well as an audio recording with information about hot flashes including treatment options.
  Arms: Self-Administered White Noise Hypnosis

SUMMARY:
The long-term goal of this program of research is to determine safe and effective non-hormonal interventions for menopausal symptoms. The main goal of this study is to evaluate whether self-administered hypnosis can be used to significantly reduce hot flashes more than self-administered white noise hypnosis over 6 weeks of home practice. The investigators are also examining the impact of each hypnosis group on sleep, anxiety, perceived and measured stress, heart rate variability, and daily activities.

DETAILED DESCRIPTION:
This randomized, two arm clinical trial will evaluate the efficacy of self-administered hypnosis for the treatment of hot flashes in postmenopausal women using a 1:1 randomization schedule.

Primary Objective

To evaluate the efficacy of the self-administered hypnosis intervention for hot flashes compared to the self-administered white noise hypnosis.

Hypothesis 1: Self-administered hypnosis will significantly decrease vasomotor symptoms (hot flash score of frequency and severity) compared to the self-administered white noise hypnosis at 6 weeks.

Secondary Objectives

To evaluate the efficacy of the self-administered hypnosis compared to self-administered white noise hypnosis for hot flash activity interference, sleep disturbance, anxiety and perception of benefit; with the expectation that there will be significant improvements among participants in the self-administered hypnosis group when compared with the self-administered white noise hypnosis group at 6 weeks. The investigators will also evaluate the effects of self-administered hypnosis compared to the self-administered white noise hypnosis at 12 weeks for all secondary outcomes except perception of benefit. Additionally, mediators (perceived stress, cortisol, and heart rate variability (HRV)) and moderators (hypnotizability and practice adherence) of hot flash reduction will be explored.

Hypothesis 2.1: Compared to self-administered white noise hypnosis, the self-administered hypnosis intervention will result in significant improvements in hot flash activity interference, sleep disturbance, and anxiety at 6 and 12 weeks, and perception of benefit at 6 weeks.

Hypothesis 2.2 A decrease in perceived stress will be indicated in the self-administered hypnosis group due to the intervention, which will correspond and contribute to further decrease of the hot flash score at 6 and 12 weeks.

Hypothesis 2.3 Diurnal salivary cortisol will demonstrate better circadian rhythms (steeper slopes) in those with larger hot flash reductions and in the self-administered hypnosis group compared to participants in the self-administered white noise hypnosis at 6 weeks.

Hypothesis 2.4 Self-administration of hypnosis and greater hot flash reductions will result in higher resting and 24-hour parasympathetic activity, reflected as higher HRV at 6 weeks.

Hypothesis 2.5 Higher hypnotizability scores and better adherence rates will be associated with greater reductions in hot flash scores in the self-administered hypnosis group.

Hypothesis 2.6 Self-administered hypnosis will significantly decrease vasomotor symptoms (hot flash score of frequency and severity) compared to the self-administered white noise hypnosis at 12 weeks.

Recruitment Plan

Potential participants will be identified in three ways: postcard mailings and invitation letters; physician referrals and IRB approved chart screening; and flyers, advertisements and press releases. Physician referrals will come primarily from cancer centers at University of Michigan Cancer Center Breast Clinic in Ann Arbor, MI, and the Baylor Scott & White Health Center in Waco, TX.

At Michigan, key eligibility criteria will be used to identify potential eligible women through the Honest Broker Office. Charts will be further screened, with IRB approval, for eligibility. If eligible, women will be sent an invitation letter where they can opt in or out of being contacted to learn more about the study.

In addition, at Michigan, outreach will occur through obstetrics and gynecology, mammography, and internal medicine clinics to enable recruitment of women without a history of breast cancer. Mass mailings and local advertisement may also be used.

At Baylor University, a successful and proven method of accrual has been the use of mass mailings and local advertisement (e.g. newspaper, magazines, flyers). Additionally, Dr. Elkins is a medical associate with Baylor Scott & White Health Center, which provides a direct connection with physicians and medical staff who will provide potential referrals.

It is expected that each site (Baylor University and University of Michigan) will recruit approximately half of the participants. Accrual will be closely monitored and efforts to randomize an equal number at each site will be made.

The study coordinators will provide education about the trial and a consent form for review both by phone and at the baseline/consent session. All other education beyond the baseline data collection will be provided at the second session 7-30 days later. Both sessions will be between 45-60 minutes. Sessions will be held at Dr. Barton's and Dr. Elkin's research offices, which each provide privacy, a recliner, a relaxing environment, and convenient parking.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal as defined by one of the following criteria:

* No menstrual period in the past 12 months
* Chemical menopause (LHRH antagonists)
* Surgical Menopause (bilateral oophorectomy)
* Evidence of menopause status per FSH and estradiol levels per institutional guidelines. Self-reported history of a minimum of 4 hot flashes per day or 28 hot flashes per week at baseline.

Age over 18 years and able to give consent for participation in the study.

Have discontinued other putative therapies for hot flashes for at least one month prior to enrollment (Vitamin E will be allowed)

Women with a diagnosis of DCIS or invasive breast cancer stages 0-III are allowed to participate and may be on endocrine therapy of any kind. If on endocrine therapy, women must be on it for 4 weeks and not expected to stop it during the study. If not on endocrine therapy, participants should not be planning to start during the course of the study. However, unexpected treatment will not require study withdrawal but will be recorded and considered in the analysis.

Exclusion Criteria:

* Currently receiving other simultaneous treatment for hot flashes (antidepressant use is allowed if being used for mood alterations and participant has been on the antidepressant for at least 3 months with no plans to change dose or antidepressant during this study)
* Diagnosis of clinical depression or acute anxiety disorder
* Currently using any Complementary and Alternative Medicine (CAM) treatments for vasomotor symptoms. (This would include soy products and other phytoestrogens, black cohosh, and any mind-body techniques including meditation, yoga, etc.). If any therapies are used for reasons other than hot flashes and hot flash frequency meets inclusion criteria, then woman is eligible)
* Diagnosis of a serious psychological illness, specifically psychoses, schizophrenia or borderline personality disorder
* Currently using hypnosis for any reason
* PHQ-4 score ≥ 9
* Non-English speaking
* Women with stage IV breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Elkins, Ph.D., Principal Investigator — Baylor University; Debra Barton, RN,PhD,FAAN, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Baylor University, Waco, Texas

REFERENCES:
- [Derived] Elkins G, Arring N, Morgan G, Lorenz T, Muniz V, Lafferty C, Scheffrahn K, Alldredge C, Barton D. Self-Administered Hypnosis vs Sham Hypnosis for Hot Flashes: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2542537. doi: 10.1001/jamanetworkopen.2025.42537. PMID 41217756

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-Administered Hypnosis | Self-Administered White Noise Hypnosis
Started | 126 | 124
Completed | 107 | 97
Not Completed | 19 | 27

BASELINE CHARACTERISTICS:
Groups:
- Self-Administered White Noise Sham Hypnosis: Self-administered white noise hypnosis will be practiced daily using a white noise recording. Participants will practice hypnosis at home after completing the two consent and education sessions.
  Self-Administered White Noise Hypnosis: Participants will be listening to the same 20-minute white noise audio recordings for 6 weeks and will be encouraged to practice daily.They will also be provided with booklets as well as an audio recording with information about hot flashes including treatment options.
- Total: Total of all reporting groups
Arm/Group | Self-Administered Hypnosis | Self-Administered White Noise Sham Hypnosis | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.69 (6.67) | 56.17 (7.17) | 55.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 124 | 250
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 118 | 115 | 233
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 20 | 39
  White | 96 | 91 | 187
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 126 | 124 | 250
Breast Cancer Survivor [Count of Participants; unit: Participants] | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Daily Diary
Description: Participants completed the Hot Flash Daily Diary (Sloan et al., 2001) every day for 6 weeks to measure the daily frequency and severity (mild, moderate, severe, and very severe) of hot flashes. A total hot flash score was calculated for each participant (product of frequency x severity) after severity ratings were assigned a point value as follows:
  * mild = 1
  * moderate = 2
  * severe = 3
  * very severe = 4 The hot flash score was then calculated by multiplying the participants' frequency and severity ratings of hot flashes, divided by the total number of days. A lower score indicates less frequent and/or severe hot flashes.
Time Frame: The hot flash daily diary was collected at baseline (week 0), endpoint (week 6) and follow-up (week 12).
Measure: Mean (Standard Deviation); unit: Hot Flash Score
Groups:
- Self-Administered Sham Hypnosis: Self-administered sham hypnosis will be practiced daily using a white noise recording. Participants will practice hypnosis at home after completing the two consent and education sessions.
  Self-Administered Sham Hypnosis: Participants will be listening to the same 20-minute white noise audio recordings for 6 weeks and will be encouraged to practice daily.They will also be provided with booklets as well as an audio recording with information about hot flashes including treatment options.
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
Hot Flash Score
  Baseline (Week 0) | 88.7 (61.3) | 94.6 (81.6)
  Endpoint (Week 6) | 41.3 (50.8) | 55.9 (50.9)
  Follow-up (Week 12) | 34.7 (34.4) | 52.8 (49.4)

2. Secondary Outcome: Hot Flash Related Daily Interference Scale
Description: This is a 10-item scale that measures hot flash interference. The Hot Flash Related Daily Interference Scale asks respondents to rate the degree on a 0 (not at all) - 10 (very much so) scale that the hot flashes interfere with various daily activities as well as overall enjoyment or quality of life. The total score will range from 0-100. The higher the total score, the more likely hot flashes are interfering with the daily activities.This measure has been shown to be valid and internally consistent with Cronbach's alpha of .96.
Time Frame: The Hot Flash Related Daily Interference Scale was completed at Baseline (week 0), at endpoint (week 6) and at follow-up (week 12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
score on a scale
  Baseline | 49.3 (22.6) | 47.3 (22.4)
  Endpoint | 25 (22.4) | 29.6 (22)
  Follow-up | 21.4 (20.2) | 24.2 (20.3)

3. Secondary Outcome: Emotional Distress Anxiety Scale
Description: This 29-item scale measures 5 domains of anxiety: 1) affective, 2)cognitive, 3) somatic, 4) behavioral, and 5) need for treatment. Items are scored on a scale from 1 (never) - 5 (always) with higher scores reflecting more severe anxiety. The total range for this scale is 0-145. This scale has shown excellent convergent and discriminate validity with other measures with a Cronbach's alpha .95.
Time Frame: Baseline, 6 & 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
units on a scale
  Baseline | 49.83 (16.19) | 50.82 (16.98)
  Endpoint | 45.93 (15.05) | 47.59 (16.74)
  Follow-up | 44.85 (16.60) | 47.79 (16.77)

4. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: This is a 19-item self-report inventory designed to measure sleep disturbance. The 19 items are grouped into 7 sub-scales: 1) sleep quality; 2) sleep efficiency; 3) daytime dysfunction; 4) sleep latency; 5) sleep disturbances; 6) sleep duration; and 7) use of sleep medication.These seven sub-scales are scored on a scale of 0 (better) - 3 (worse) with higher scores indicating greater sleep pathology. The sub-scales are then added for a combined total score ranging from 0 (better) - 21 (worse). Alphas for the Pittsburgh Sleep Quality Index range from .70 to .80.
Time Frame: Baseline, 6, & 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
units on a scale
  Baseline | 7.08 (2.23) | 7.13 (2.51)
  Endpoint | 6.23 (2.53) | 6.31 (2.39)
  Follow-up | 6.33 (2.31) | 6.10 (2.15)

5. Secondary Outcome: Subject Global Impression of Change
Description: Participants were asked to fill out the Subject Global Impressions of Change at endpoint (week 6) to gauge participants' perceived benefit. The Subject Global Impression of Change is a single item in which the participant rates, from 0 to 4, the change in hot flashes since beginning the study. Response options range from "not at all" (0), "a little" (1), "somewhat" (2), "quite a bit" (3), "totally satisfied" (4). The question used was, "How satisfied are you with the impact of the study treatment on your hot flashes?". This question has been used extensively for determination of minimally clinically significant differences in numerous oncology clinical trials prior to this study.
Time Frame: The Subject Global Impressions of Change will be completed only at 6 weeks.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
Units on a Scale | 1.92 (1.066) | 1.20 (1.228)

6. Secondary Outcome: Perceived Stress Scale
Description: This is a 10-item scale that measures the degree to which situations in one's life are appraised as stressful. The scale provides the degree to which individuals find their lives to be unpredictable, uncontrollable, and overloaded, as well as measures the current levels of experienced stress. Items are scored on a scale from 0 (never) - 4(very often) for a total score ranging from 0-40. with higher scores reflecting more perceived stress. This measure has been shown to be valid and internally consistent, with an alpha of .83.
Time Frame: Baseline, 6, & 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
units on a scale
  Baseline | 12.38 (6.686) | 12.11 (6.647)
  Week 6 | 11.36 (6.368) | 11.16 (6.874)
  Week 12 | 10.26 (6.123) | 10.64 (6.935)

7. Other Pre Specified Outcome: Self-Hypnosis Practice Log
Description: Participants in both groups were given the Self-Hypnosis Practice Log to record daily practice of self-hypnosis or sham hypnosis throughout the 6-week intervention period and at the week 12 follow-up as a measure of intervention adherence. Adherence scores (number of practices per week) were calculated as the total frequency of reported practices according to group assignment in a seven-day period with or without the aid of an audio recording. Average adherence was calculated by averaging the adherence scores of week 1(initiation of study), week 6 (end of intervention), and week 12 (follow-up).
Time Frame: The practice log was completed daily by the participants and submitted to the interventionists at the end of each week throughout the study's duration (weeks one through six) and at follow-up (week 12)."
Measure: Mean (Standard Deviation); unit: Number of practices per week
Arm/Group | Self-Administered Hypnosis | Self-Administered Sham Hypnosis
Number analyzed (Participants) | 126 | 124
Number of practices per week
  Baseline | 7.4 (4.4) | 7.6 (3.4)
  Endpoint | 10.9 (6.6) | 7.4 (3.1)
  Follow-up | 8.3 (7.2) | 5.6 (5.1)

ADVERSE EVENTS:
Time Frame: All participants were monitored for Adverse Events during the entire study duration, an average of 3 months.
Description: Any serious adverse events were reported to the IRB and NCCIH.
Groups:
- Intervention: Self-Administered Hypnosis
- Control: Self-Administered Sham Hypnosis
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/124
Other Adverse Events (participants affected / at risk) | 4/126 | 5/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=126) | Control (N=124)
Mild/Moderate Adverse Events (General disorders) | 4 (7) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT03572153/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03572153/ICF_001.pdf